CLINICAL TRIAL: NCT05692427
Title: Evaluation of Cryotherapy in Granuloma Pyogenicum by Means of Cryopen Compared to Surgical Removal
Brief Title: Evaluation of Cryotherapy in Granuloma Pyogenicum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 34-028 ex 21/22
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Granuloma, Pyogenic; Cryotherapy Effect
MeSH Terms: conditions — Granuloma, Pyogenic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryotherapy (Other): Cryotherapy on granuloma pyogenicum
  Interventions: Device: Cryopen - Cryotherapy

INTERVENTIONS:
Device: Cryopen - Cryotherapy — Cryotherapy with N20

SUMMARY:
Surgical excision needs general anesthesia and might have complications due to anesthesia. Cryotherapy can be used in an outpatient setting and doesn't need general anesthesia.

This study will evaluate if cryotherapy works in granuloma pyogenicum with the advancement of no general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

diagnosis of granuloma pyogenicum

Exclusion Criteria:

no approvement of cryotherapy

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Granuloma pyogenicum | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided